CLINICAL TRIAL: NCT03254680
Title: Turmeric as Treatment in Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00750
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Epilepsy; Dravet Syndrome; Lennox-Gastaut Syndrome; Tuberous Sclerosis; Focal Seizures
Keywords: Turmeric Oil; antiseizure medications; ar-turmerone
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Lennox Gastaut Syndrome; Tuberous Sclerosis; Seizures | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Turmeric Oil (Experimental): stable dose of orally administered turmeric oil
  Interventions: Dietary Supplement: Turmeric

INTERVENTIONS:
Dietary Supplement: Turmeric — Twenty patients will be enrolled and treated with a stable dose of orally administered turmeric oil daily for 3 months.

SUMMARY:
This is a single center open-label pilot clinical trial of patients 1-70 years of age with greater than 6 seizures per month diagnosed with Dravet Syndrome, Lennox-Gastaut Syndrome, Tuberous Sclerosis, or focal seizures. Twenty patients will be enrolled and treated with a stable dose of orally administered turmeric oil daily for 3 months. Patients and caregivers will be asked to keep a seizure diary logging all clinical events during the course of the study. Serum comprehensive metabolic panel, complete blood count with differential, and antiseizure medication levels, will be monitored at baseline, 1.5 months, and at the end of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with greater than greater than six seizures per month diagnosed with Dravet Syndrome, Lennox-Gastaut Syndrome, Tuberous Sclerosis, or focal seizures followed at NYU CEC.

Exclusion Criteria:

* Patients expected to have changes to any medications or supplements during study period
* exposure to any investigational agent in the month prior to study entry
* pregnant or breast feeding women, positive pregnancy test
* history of non-compliance
* known drug or alcohol dependence
* known baseline hematologic
* liver function
* renal function
* absorption
* absorption

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Number of epilepsy patients enrolled in study | 3 months
  feasibility of recruiting patients into a prospective study designed to evaluate the effect of orally ingested turmeric oil on seizures.

SECONDARY OUTCOMES:
Number of epilepsy seizures post epilepsy treatment with turmeric | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Holmes, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided